CLINICAL TRIAL: NCT05972928
Title: Effect of Sitagliptin on Clinical, Metabolic and Hormonal Parameters in Polycystic Ovarian Syndrome Patients
Brief Title: Effect of Sitagliptin on Polycystic Ovarian Syndrome Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sitagliptin PCO
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Sitagliptin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin at a dose of 100 mg every 24 hours for 3 months
  Interventions: Drug: Sitagliptin 100mg
- control (No Intervention): patient won't receive medication

INTERVENTIONS:
Drug: Sitagliptin 100mg — Sitagliptin at a dose of 100 mg every 24 hours for 3 months
  Other Names: Januvia 100 mg tab
  Arms: Sitagliptin

SUMMARY:
The Study aims to determine the proposed positive influence of Sitagliptin in manipulating hormonal , metabolic and inflammatory parameters in the treatment of Polycystic ovary syndrome and subsequent infertility

DETAILED DESCRIPTION:
Study Design : a Prospective Randomized Controlled Trial.

A Total of 80 infertile Adult Females aged between 18 and 45 years currently diagnosed with Polycystic ovary syndrome , Meeting the Diagnosis of Rotterdam criteria be diagnosed if any two of the following are present: (1) clinical or biochemical hyperandrogenism, (2) evidence of oligo-anovulation, (3) polycystic appearing-ovarian morphology on ultrasound are to be included in the study.

The study will include two groups; each group consists of 40 patients:- Group A : Control Group Group B : Test Group ( will Receive Sitagliptin at a dose of 100 mg every 24 hours

ELIGIBILITY:
Inclusion Criteria:

polycystic ovary syndrome usually diagnosed based on the Rotterdam criteria if 2 of 3 criteria are present:

1. oligo- and/or anovulation
2. hyperandrogenism (HA) (clinical and/or biochemical)
3. polycystic ovary morphology (PCOM) on ultrasonography (either 12 or more follicles measuring 2-9 mm in diameter and/or an increased ovarian volume >10 cm3).

Exclusion Criteria:

1. congenital adrenal hyperplasia
2. Brittle control of a thyroid disorder
3. Diabetic on Metformin or any another antidiabetic drugs affecting insulin resistance
4. chronic kidney disease
5. liver dysfunction
6. documented use of oral hormonal contraceptives and hormone-releasing implants in the past 6 months prior to study entry 7.Lipid lowering Consumption

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Body weight loss in Kilograms | 3 months
  Body weight before - Body weight after

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided